CLINICAL TRIAL: NCT01194804
Title: Phase II Clinical Study of Eculizumab (h5G1.1-mAb) in Hemolytic Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients: Extension Study to C07-001 Protocol
Brief Title: E07-001: Safety and Efficacy Extension Study of Eculizumab in Paroxysmal Nocturnal Hemoglobinuria Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: CMIC Co, Ltd. Japan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E07-001
Record Dates: First submitted 2010-08-30; First posted 2010-09-03 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: Hemolytic Paroxysmal Nocturnal Hemoglobinuria; Eculizumab; PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eculizumab (Experimental): Treatment with eculizumab for patients with PNH who have successfully completed the C07-001 protocol
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Each vial contains 30 mL of 10 mg/mL eculizumab; dose of 900 mg intravenous every 14 days.
  Other Names: Soliris

SUMMARY:
The objective of this study was to assess the long-term safety and efficacy of eculizumab in hemolytic PNH patients who completed the 4-week screening and 12-week treatment period of the C07-001 study. In addition, pharmacokinetic and pharmacodynamic assessments of eculizumab were conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have fully completed C07-001 study 12-week treatment period

Exclusion Criteria:

* Patients who terminated early from the C07-001 study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kanakura Y, Ohyashiki K, Shichishima T, Okamoto S, Ando K, Ninomiya H, Kawaguchi T, Nakao S, Nakakuma H, Nishimura J, Kinoshita T, Bedrosian CL, Ozawa K, Omine M. Long-term efficacy and safety of eculizumab in Japanese patients with PNH: AEGIS trial. Int J Hematol. 2013 Oct;98(4):406-16. doi: 10.1007/s12185-013-1404-y. Epub 2013 Aug 11. PMID 23934275

RESULTS

PARTICIPANT FLOW:
Groups:
- Eculizumab: Treatment with eculizumab for patients with paroxysmal nocturnal hemoglobinuria who have successfully completed the C07-001 protocol (NCT01192399)
  Eculizumab: 900 mg intravenous every 14 days.
Period: Overall Study
Arm/Group | Eculizumab
Started | 27
Completed | 26
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Eculizumab: Treatment with eculizumab for patients with PNH who have successfully completed the C07-001 protocol
  900 mg intravenous every 14 days.
Arm/Group | Eculizumab
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (12.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 27
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 27

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lactate Dehydrogenase
Time Frame: 52 weeks (includes 12 weeks of eculizumab treatment in the parent study and 40 weeks in the extension study)
Measure: Mean (Standard Error); unit: Units/Liter
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
Units/Liter | -15.9 (1.20)
Statistical Analysis 1: Comparison: Eculizumab; Test type: Other; p < 0.001, Sign test

2. Secondary Outcome: Change From Baseline in FACIT-Fatigue Scale Total Score
Description: The FACIT-Fatigue scale, Version 4.0, is a collection of quality of life questionnaires pertaining to the management of fatigue symptoms due to a chronic illness. The FACIT-Fatigue is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the preceding 7 days. Patients score each item on a 5-point scale: 0 (Not at all) to 4 (Very much). Total scores range from 0 to 52, with higher score indicating better quality of life.
Time Frame: 52 weeks (includes 12 weeks of eculizumab treatment in the parent study and 40 weeks in the extension study)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
units on a scale | 8.0 (1.95)

3. Secondary Outcome: Change From Baseline in PNH Red Blood Cell (RBC) Count
Time Frame: 52 weeks (includes 12 weeks of eculizumab treatment in the parent study and 40 weeks in the extension study)
Measure: Mean (Standard Error); unit: cellsx10^12/L
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
cellsx10^12/L | 0.51 (0.129)

4. Secondary Outcome: Change From Baseline in Number of Units of Packed RBCs Transfused
Description: Baseline is defined as the number of units transfused in 3 months prior to baseline
Time Frame: 52 weeks (includes 12 weeks of eculizumab treatment in the parent study and 40 weeks in the extension study)
Measure: Mean (Standard Error); unit: units
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
units | -3.5 (1.43)

5. Secondary Outcome: Change From Baseline in Plasma Free Hemoglobin
Time Frame: 52 weeks (includes 12 weeks of eculizumab treatment in the parent study and 40 weeks in the extension study)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Eculizumab
Number analyzed (Participants) | 26
mg/dL | -13.5 (8.55)

ADVERSE EVENTS:
Time Frame: From baseline (after first dose) to end of study (1 year).
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 12/27
Other Adverse Events (participants affected / at risk) | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=27)
Anaemia (Blood and lymphatic system disorders) | 2
Haemolysis (Blood and lymphatic system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 4
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=27)
Anaemia (Blood and lymphatic system disorders) | 3
Conjunctival haemorrhage (Eye disorders) | 3
Cataract (Eye disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Abdominal discomfort (Gastrointestinal disorders) | 2
Dental caries (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 2
Mouth ulceration (Gastrointestinal disorders) | 2
Pyrexia (General disorders) | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 2
Nasopharyngitis (Infections and infestations) | 21
Upper respiratory tract infection (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 3
Laceration (Injury, poisoning and procedural complications) | 2
Blood alkaline phosphatase increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 6
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes